CLINICAL TRIAL: NCT05783492
Title: Intranasal Ketamine for Procedural Sedation: a Feasibility Cohort Study
Brief Title: INK Feasibility Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of availability of drug
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113103
Record Dates: First submitted 2018-11-23; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2018-11

CONDITIONS: Procedural Sedation
Keywords: ketamine

STUDY DESIGN:
Intervention Model Description: Intranasal ketamine 10 mg/kg single dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intranasal ketamine (Experimental): Intranasal ketamine 10 mg/kg
  Interventions: Drug: Intranasal ketamine

INTERVENTIONS:
Drug: Intranasal ketamine — 10 mg/kg single dose in 0.5 mL sprays in each nare separated by 60 seconds

SUMMARY:
The trial (Intranasal ketamine for procedural sedation in children: a randomized controlled non-inferiority multicenter trial or INK; ReDA 5496; CTO 1545) is being scheduled for launch in Spring 2019. Due to the possibility of failure of the experimental intervention (intranasal ketamine 10 mg/kg), the data safety monitoring board (DSMB) and statistical methods team would like to explore the possibility of developing a stopping rule to prevent patients from being enrolled in a futile trial and conserve resources. In order to get accurate data to develop a statistically robust stopping rule, it is necessary to conduct a cohort study of patients that receive the INK trial's experimental intervention and according to it's protocol. This cohort study will help estimate the chance of adequate sedation and inform the final dosing protocol for the INK trial.

DETAILED DESCRIPTION:
Between 20 and 40% of extremity fractures in children require a closed reduction, often necessitating procedural sedation and analgesia (PSA) (3, 4). Intravenous (IV) ketamine is the most commonly used sedative agent used to perform a closed reduction (5). However, children rate IV insertion as the most painful hospital experience, second only to the injury itself (6). Intranasal (IN) ketamine may provide effective sedation for children undergoing a closed reduction without the distress and pain related to IV insertion. Although the proportion of children with adequate sedation using IN ketamine at doses of 9-10 mg/kg has been reported to be at least 75% (9-11), there is the possibility of inadequate sedation because IN ketamine 10 mg/kg has not been used for procedural sedation for fracture reduction. A multi-centre, two-arm, randomized, blinded, controlled, non-inferiority trial designed to test the hypothesis that intranasal (IN) ketamine is non-inferior to intravenous (IV) ketamine is being planned for launch in Spring 2019 and a stopping rule for futility will ensure that patients are not unduly enrolled and that resources are not wasted in a futile trial. Creating of a methodologically rigorous stopping rule depends on the results of a small cohort study to provide a more accurate and informed estimate of the probability of adequate sedation with IN ketamine 10 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* General Criteria

  1. Provision of signed and dated informed consent form
  2. Stated willingness to comply with all study procedures and availability for the duration of the study
  3. Deemed by treating physician to require procedural sedation using ketamine Specific Criteria

  <!-- -->

  1. Children presenting to the paediatric EDs of participating sites age 7-17 years
  2. Weighing up to and including 80 kg
  3. Distal radius +/- ulna fracture or dislocation of a shoulder, elbow, patella, or digit
  4. Closed reduction expected to take no more than 5 minutes to reduce (as determined by the procedure physician and not including cast or splint application).

Exclusion Criteria:

* 1) Previous hypersensitivity reaction to ketamine including rash, difficulty breathing, hypotension, apnea, or laryngospasm; 2) Suspected globe rupture; 3) Concomitant traumatic brain injury with intracranial hemorrhage; 4) Uncontrolled hypertension; 5) Nasal bone deformity or nasal obstruction with at least one nare obstructed due to allergic or viral rhinitis, sinusitis, nasal polyps, or septal deviation; 6) Poor English or French fluency in the absence of native language interpreter; 7) American Society of Anesthesiologists (ASA) class 3 or greater; 8) Previous diagnosis of schizophrenia or active psychosis as per the treating physician 9) Neuro-cognitive impairment that precludes informed consent, assent, or ability to self-report pain and satisfaction; 10) Multi-limb trauma; 11) Hemodynamic compromise as per the treating physician; 12) Glasgow coma score < 15; 13) Previous sedation with ketamine within 24 hours; 14) Fracture is comminuted or associated with a dislocation; 15) Participant has undergone a hematoma block within 24 hours; 16) Isolated ulna fracture; 17) Previous enrollment in the trial; 18) Suspected pregnancy

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Adequacy of sedation | 1 hour
  Dartmouth Operative Conditions Scale (DOCS) score between -2 and +2 for the duration of the closed reduction AND, (ii) No additional IV ketamine is given during closed reduction for the purpose of sedation, AND (iii) The patient did not actively resist, cry, or require physical restraint for completion of the closed reduction.

SECONDARY OUTCOMES:
Length of stay | 1 hour
  Defined as the time recorded in the medical record between triage and discharge in minutes
Onset of sedation | 1 hour
  This will be defined as the time interval from administration of the first pair of IN sprays to the time when a first DOCS score of between -2 and +2 is achieved post-intervention (minutes)
Duration of sedation | 1 hour
  This will be defined as the duration of time between the first DOCS score between -2 to +2 post-intervention to the last DOCS score between -2 and +2 post-closed reduction (minutes).
Adverse effects | 1 hour
  Research nurses will be trained on the recognition and definition of expected and unexpected AEs. AEs will be determined from the medical record and recorded on REDCap. Expected AEs are based on the Quebec guidelines and other practice guidelines. Unpleasant recovery reactions will be recorded by the research nurse using REDCap.

IPD SHARING:
Plan to Share IPD: No